CLINICAL TRIAL: NCT07014358
Title: Randomized, Patient-blinded, Evaluator-blinded Clinical Trial With Three CE-marked and Approved Devices
Brief Title: Clinical Trial to Evaluate Three Systems of Osteosynthesis for Fixation of Olecranon Osteotomies in Adults
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIJAOLE01
Record Dates: First submitted 2025-05-13; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Olecranon Fracture
MeSH Terms: conditions — Olecranon Fracture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fastening systems by placing two steel pins (Experimental): Fixation of the osteotomized bone with a stable fixation system, in this case, the placement of two steel pins.
  Interventions: Device: Fastening systems by placing two steel pins
- Fastening systems by a wire in an obenque configuration (Experimental): Fixation of the osteotomized bone with a stable fixation system, in this case, an obenque configuration.
  Interventions: Device: Fastening systems by a wire in an obenque configuration
- Fastening systems by the placement of a bolted plate or the placement of a compression screw (Experimental): Fixation of the osteotomized bone with a stable fixation system, in this case, the placement of a bolted plate or the placement of a compression screw.
  Interventions: Device: Fastening systems by the placement of a bolted plate or the placement of a compression screw

INTERVENTIONS:
Device: Fastening systems by placing two steel pins — Fixation of the osteotomized bone with a stable fixation system, in this case, the placement of two steel pins.
  Arms: Fastening systems by placing two steel pins
Device: Fastening systems by a wire in an obenque configuration — Fixation of the osteotomized bone with a stable fixation system, in this case, an obenque configuration
  Arms: Fastening systems by a wire in an obenque configuration
Device: Fastening systems by the placement of a bolted plate or the placement of a compression screw — Fixation of the osteotomized bone with a stable fixation system, in this case, the placement of a bolted plate or the placement of a compression screw.
  Arms: Fastening systems by the placement of a bolted plate or the placement of a compression screw

SUMMARY:
Surgery of the elbow joint is often made difficult by the highly constrained nature of the elbow joint. This is why it is often necessary to perform an osteotomy of the olecranon, the proximal part of the ulna, which allows perfect exposure of the entire articular surface. After performing the osteotomy, access to the joint is obtained, the articular problem is solved as appropriate and, upon completion, the osteotomized bone is fixed with a stable fixation system that allows the osteotomy to heal without problems. It is a safe, reproducible procedure that is associated with low associated morbidity. The main problems associated with this procedure are the lack of consolidation of the osteotomy or the need for removal of the osteosynthesis material at a later stage.

DETAILED DESCRIPTION:
The incidence of these complications is around 4% for the former and 20-50% for the latter. Both complications usually require a second surgical procedure to solve the problem, so the reoperation rates for these procedures are around 40-50%.

However, there is discussion in the literature as to the most appropriate fixation system to ensure fracture healing. There are, broadly speaking, three frequently used fixation systems: the placement of two steel pins and a wire in an obenque configuration, the placement of a screwed plate or the placement of a compression screw.

It is not clear which is the best fixation system among these three. Biomechanical studies suggest that, from this point of view, all three procedures are adequate. The choice of which is ideal should therefore be based on the ease of use and the complications associated with the procedure, in particular the reoperation rate.There are no clinical trials in the literature comparing these three fixation techniques, so there is a clear lack of knowledge in this field.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, after receiving information about the design, the purposes of the study, the possible risks that may arise from it and the fact that they may refuse to collaborate at any time, give their written consent to participate in the study.
* Be over 18 years of ag
* Have an elbow disorder that is to be treated surgically through an olecranon osteotomy approach.
* That the olecranon osteotomy is amenable to synthesization with the three proposed systems.
* Understand the purpose of the study and be available for routine hospital visits.

Exclusion Criteria:

* Patients who have undergone ipsilateral elbow surgery.
* Presence of ulnar fractures
* Patients with an active infection at any site at the time of elbow surgery.
* Inability to understand the procedure or information related to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Define which of the three fixarion systems is safer based on the number of patients with each fixation system that need to be reintervened. | 12 Months
  The main evaluation criterion will be the need for reoperation for any cause related to the olecranon osteotomy in the first year of follow-up.

SECONDARY OUTCOMES:
Number of patients suffering Adverse Events related or not with the medical product within a year | 12 months
  Infection
Number of patients suffering Adverse Events related or not with the medical product within a year | 12 months
  Complications in the healing process of the surgical wound
Number of patients suffering: Adverse Events related or not with the medical product within a year | 12 months
  Mechanical complications with the implant
Number of patients suffering Adverse Events related or not with the medical product, within a year | 12 months
  Reintervention
Number of patients suffering Adverse Events, related or not with the medical product, within a year | 12 months
  Residual pain
Number of patients suffering Adverse Events related or not, with the medical product, within a year | 12 months
  Fracture
Efficacy measured usimg the evaluation of different scales and tests performed by the patient, that altogether provide the needed information about the efficacy of the medical product. | 24 months
  Measured by Pain leveld (BPI test)
Efficacy, measured usimg the evaluation of different scales and tests performed by the patient that altogether provide the needed information about the efficacy of the medical product. | 24 months
  Measured by Mayo Elbow Score Scale (MEPS)
Efficacy, measured usimg the evaluation of different scales and tests performed by the patient, that altogether provide the needed information about the efficacy of the medical product | 24 months
  Measured by pasive and active movility range

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Mutua Montañesa Santander, Santander, Cantabria
  - Clínica CEMTRO, Madrid, Madrid
  - Hospital de Manises, Valencia, Manises
  - Hospital La Fe, Valencia, Valencia
  - Hospital Universitario de Móstoles, Madrid